CLINICAL TRIAL: NCT00847613
Title: Phase 3 Randomized, Double Blind, Placebo Controlled Study Of The Efficacy And Safety Of 2 Doses Of CP-690,550 In Patients With Active Rheumatoid Arthritis On Background Methotrexate
Brief Title: A 2-Year Phase 3 Study Of CP-690,550 In Patients With Active Rheumatoid Arthritis On Background Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921044
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: double-blind placebo-controlled investigational drug oral therapy safety and efficacy hand and feet x-rays
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sequence 1 (Experimental)
  Interventions: Drug: CP-690,550
- Sequence 2 (Experimental)
  Interventions: Drug: CP-690,550
- Sequence 3 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: CP-690,550
- Sequence 4 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — Oral tablets administered at 5 mg BID daily for 6 months (nonresponders advance to second intervention at 3 months) during the double-blind, placebo-controlled period.
  Other Names: Double-blind, placebo-controlled period
  Arms: Sequence 1
Drug: CP-690,550 — Oral tablets administered at 5 mg BID daily through the end of the study during the double-blind, active-extension period.
  Other Names: Double-blind, Active Extension Period
  Arms: Sequence 1
Drug: CP-690,550 — Oral tablets administered at 10 mg BID daily for 6 months (nonresponders advance to second intervention at 3 months) during the double-blind, placebo-controlled period.
  Other Names: Double-blind, placebo-controlled period
  Arms: Sequence 2
Drug: CP-690,550 — Oral tablets administered at 10 mg BID daily through the end of the study during the double-blind, active-extension period.
  Other Names: Double-blind, Active Extension Period
  Arms: Sequence 2
Drug: Placebo — Oral placebo tablets administered BID daily for 6 months (nonresponders advance to second intervention at 3 months) during the double-blind, placebo-controlled period.
  Other Names: Double-blind, placebo-controlled period
  Arms: Sequence 3
Drug: CP-690,550 — Oral tablets administered at 5 mg BID daily through the end of the study during the double-blind, active-extension period.
  Other Names: Double-blind, Active Extension Period
  Arms: Sequence 3
Drug: Placebo — Oral placebo tablets administered BID daily for 6 months (nonresponders advance to second intervention at 3 months) during the double-blind, placebo-controlled period.
  Other Names: Double-blind, Active Extension Period
  Arms: Sequence 4
Drug: CP-690,550 — Oral tablets administered at 10 mg BID daily through the end of the study during the double-blind, active-extension period.
  Other Names: Double-blind, placebo-controlled period
  Arms: Sequence 4

SUMMARY:
This study is designed to provide safety and efficacy data to support the development of CP-690,550 in patients with moderate to severe rheumatoid arthritis on background of methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Adults with moderate to severe rheumatoid arthritis on a stable dose of methotrexate

Exclusion Criteria:

* Pregnancy, severe acute or chronic medical conditions, including serious infections or clinically significant laboratory abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (100):
- United States (35):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Maria, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Morton Grove, Illinois
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Lee's Summit, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Binghamton, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Clarksburg, West Virginia
  - Pfizer Investigational Site, Franklin, Wisconsin
- Australia (3):
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Woodville, South Australia
  - Pfizer Investigational Site, Malvern East, Victoria
- Brazil (5):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (2):
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Sofia
- Canada (8):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Colombia (4):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Bucaramanga, Santander Department
- Czechia (7):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Brno-Židenice
  - Pfizer Investigational Site, Hostivice
  - Pfizer Investigational Site, Pardubice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 11 - Chodov
  - Pfizer Investigational Site, Zlín
- Pfizer Investigational Site, Thessaloniki, Greece
- India (5):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Secunderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Pune, Maharashtra
- Japan (13):
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Higashihiroshima, Hiroshima
  - Pfizer Investigational Site, Hitachi-shi, Ibaraki
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Koushi, Kumamoto
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Ohmura, Nagasaki
  - Pfizer Investigational Site, Sasebo, Nagasaki
  - Pfizer Investigational Site, Ureshino-shi, Saga-ken
  - Pfizer Investigational Site, Kawagoe-shi, Saitama
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Morelia, Michoacán
- Poland (2):
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- South Korea (3):
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
- Taiwan (5):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Kweishan, Taoyuan County
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Ukraine (5):
  - Pfizer Investigational Site, Simferopol, Autonomous Republic of Crimea
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Vinnitsa

REFERENCES:
- [Derived] Strand V, Schulze-Koops H, Al-Emadi S, Kinch CD, Gruben D, Germino R, Connell CA, Mysler E. Sex differences in the efficacy, safety and persistence of tofacitinib in patients with rheumatoid arthritis: a post hoc analysis of phase III and long-term extension trials. BMJ Open. 2025 Dec 24;15(12):e082366. doi: 10.1136/bmjopen-2023-082366. PMID 41448717
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Citera G, Jain R, Irazoque F, Madariaga H, Gruben D, Wang L, Stockert L, Santana K, Ebrahim A, Ponce de Leon D. Tofacitinib Efficacy in Patients with Rheumatoid Arthritis and Probable Depression/Anxiety: Post Hoc Analysis of Phase 3 and 3b/4 Randomized Controlled Trials. Rheumatol Ther. 2024 Feb;11(1):35-50. doi: 10.1007/s40744-023-00612-7. Epub 2023 Nov 5. PMID 37925660
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Dikranian AH, Gonzalez-Gay MA, Wellborne F, Alvaro-Gracia JM, Takiya L, Stockert L, Paulissen J, Shi H, Tatulych S, Curtis JR. Efficacy of tofacitinib in patients with rheumatoid arthritis stratified by baseline body mass index: an analysis of pooled data from phase 3 studies. RMD Open. 2022 May;8(1):e002103. doi: 10.1136/rmdopen-2021-002103. PMID 35577477
- [Derived] Bartlett SJ, Bingham CO, van Vollenhoven R, Murray C, Gruben D, Gold DA, Cella D. The impact of tofacitinib on fatigue, sleep, and health-related quality of life in patients with rheumatoid arthritis: a post hoc analysis of data from Phase 3 trials. Arthritis Res Ther. 2022 Apr 5;24(1):83. doi: 10.1186/s13075-022-02724-x. PMID 35382883
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Strand V, Kaine J, Alten R, Wallenstein G, Diehl A, Shi H, Germino R, Murray CW. Associations between Patient Global Assessment scores and pain, physical function, and fatigue in rheumatoid arthritis: a post hoc analysis of data from phase 3 trials of tofacitinib. Arthritis Res Ther. 2020 Oct 15;22(1):243. doi: 10.1186/s13075-020-02324-7. PMID 33059710
- [Derived] van der Heijde D, Landewe RBM, Wollenhaupt J, Strengholt S, Terry K, Kwok K, Wang L, Cohen S. Assessment of radiographic progression in patients with rheumatoid arthritis treated with tofacitinib in long-term studies. Rheumatology (Oxford). 2021 Apr 6;60(4):1708-1716. doi: 10.1093/rheumatology/keaa476. PMID 33057725
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] van der Heijde D, Strand V, Tanaka Y, Keystone E, Kremer J, Zerbini CAF, Cardiel MH, Cohen S, Nash P, Song YW, Tegzova D, Gruben D, Wallenstein G, Connell CA, Fleischmann R; ORAL Scan Investigators. Tofacitinib in Combination With Methotrexate in Patients With Rheumatoid Arthritis: Clinical Efficacy, Radiographic, and Safety Outcomes From a Twenty-Four-Month, Phase III Study. Arthritis Rheumatol. 2019 Jun;71(6):878-891. doi: 10.1002/art.40803. Epub 2019 Apr 24. PMID 30666826
- [Derived] Kivitz AJ, Cohen S, Keystone E, van Vollenhoven RF, Haraoui B, Kaine J, Fan H, Connell CA, Bananis E, Takiya L, Fleischmann R. A pooled analysis of the safety of tofacitinib as monotherapy or in combination with background conventional synthetic disease-modifying antirheumatic drugs in a Phase 3 rheumatoid arthritis population. Semin Arthritis Rheum. 2018 Dec;48(3):406-415. doi: 10.1016/j.semarthrit.2018.07.006. Epub 2018 Jul 19. PMID 30177460
- [Derived] Hall S, Nash P, Rischmueller M, Bossingham D, Bird P, Cook N, Witcombe D, Soma K, Kwok K, Thirunavukkarasu K. Tofacitinib, an Oral Janus Kinase Inhibitor: Pooled Efficacy and Safety Analyses in an Australian Rheumatoid Arthritis Population. Rheumatol Ther. 2018 Dec;5(2):383-401. doi: 10.1007/s40744-018-0118-2. Epub 2018 Jun 11. PMID 29949132
- [Derived] Strand V, Kavanaugh A, Kivitz AJ, van der Heijde D, Kwok K, Akylbekova E, Soonasra A, Snyder M, Connell C, Bananis E, Smolen JS. Long-Term Radiographic and Patient-Reported Outcomes in Patients with Rheumatoid Arthritis Treated with Tofacitinib: ORAL Start and ORAL Scan Post-hoc Analyses. Rheumatol Ther. 2018 Dec;5(2):341-353. doi: 10.1007/s40744-018-0113-7. Epub 2018 May 14. PMID 29761420
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] van der Heijde D, Tanaka Y, Fleischmann R, Keystone E, Kremer J, Zerbini C, Cardiel MH, Cohen S, Nash P, Song YW, Tegzova D, Wyman BT, Gruben D, Benda B, Wallenstein G, Krishnaswami S, Zwillich SH, Bradley JD, Connell CA; ORAL Scan Investigators. Tofacitinib (CP-690,550) in patients with rheumatoid arthritis receiving methotrexate: twelve-month data from a twenty-four-month phase III randomized radiographic study. Arthritis Rheum. 2013 Mar;65(3):559-70. doi: 10.1002/art.37816. PMID 23348607
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921044&StudyName=A%202-Year%20Phase%203%20Study%20Of%20CP-690%2C550%20In%20Patients%20With%20Active%20Rheumatoid%20Arthritis%20On%20Background%20Methotrexate

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg: CP-690,550 5 milligram (mg) tablet orally twice daily up to Month 24.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Month 24.
- Placebo, Then CP-690,550 5 mg: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20 percent (%) reduction from baseline in both swollen and tender joint counts, received CP-690,550 5 mg tablet orally twice daily up to Month 24. At Month 6, remaining participants received CP-690,550 5 mg tablet orally twice daily up to Month 24.
- Placebo, Then CP-690,550 10 mg: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction from baseline in both swollen and tender joint counts, received CP-690,550 10 mg tablet orally twice daily up to Month 24. At Month 6, remaining participants received CP-690,550 10 mg tablet orally twice daily up to Month 24.
Period: Overall Study
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Started | 321 | 319 | 81 | 79
Treated | 321 | 316 | 81 | 79
Completed | 0 | 0 | 0 | 0
Not Completed | 321 | 319 | 81 | 79
Not completed — Ongoing at cut-off date | 250 | 265 | 64 | 64
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Adverse Event | 36 | 26 | 5 | 6
Not completed — Lack of Efficacy | 7 | 3 | 3 | 1
Not completed — Study terminated by Sponsor | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 5 | 0 | 0 | 3
Not completed — Protocol Violation | 6 | 6 | 3 | 1
Not completed — Pregnancy | 1 | 1 | 0 | 0
Not completed — Site closure | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 11 | 2 | 2
Not completed — Participant moved | 4 | 1 | 0 | 0
Not completed — Sponsor request | 0 | 1 | 0 | 0
Not completed — Randomized, but not treated | 0 | 3 | 0 | 0
Not completed — Other | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Total
Number analyzed (Participants) | 321 | 316 | 81 | 79 | 797
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.6) | 52.0 (11.4) | 53.2 (11.5) | 52.1 (11.8) | 52.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 273 | 65 | 72 | 679
  Male | 52 | 43 | 16 | 7 | 118

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 6
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 6 analysis.
Time Frame: Month 6
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure. Missing values due to withdrawal or advancement to active treatment before Month 6 were imputed using Non-responder Imputation (NRI) method.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction from baseline in both swollen and tender joint counts, received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 24. At Month 6, remaining participants received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 24.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 309 | 309 | 154
percentage of participants | 51.46 | 61.81 | 25.32
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of each dose of CP-690,550 to placebo; Test type: Superiority or Other; p < 0.0001, Normal approximation — A step-down procedure was used to control for multiple comparisons. In order for the comparison to 5 mg to be statistically significant, the comparison to 10 mg had to be statistically significant; Percent difference = 36.48, 95% CI 2-sided [27.73 to 45.23]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Normal approximation — [p-value comment as in outcome 1, analysis 1]; Percent difference = 26.13, 95% CI 2-sided [17.28 to 34.97]

2. Primary Outcome: Changes From Baseline in Modified Total Sharp Score (mTSS) at Month 6
Description: mTSS = sum of erosion and Joint Space Narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change: scores at observation minus score at baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 6 analysis.
Time Frame: Baseline, Month 6
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 286 | 295 | 139
units on a scale
  Baseline | 28.66 (2.98) | 34.66 (2.95) | 29.53 (4.25)
  Change at Month 6 | 0.12 (0.12) | 0.06 (0.11) | 0.47 (0.16)
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Change at Month 6: Linear mixed model with treatment effect and site location as fixed effects and baseline value as covariate was used for the analysis; Test type: Superiority or Other; p = 0.0376, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For comparison of 10 mg to placebo to be statistically significant in this measure, comparison of 10 mg to placebo in ACR20 had to be significant; Least squares mean difference = -0.40, 95% CI 2-sided [-0.79 to -0.02], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0792, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For comparison of 5 mg to placebo to be statistically significant, comparison of 10 mg to placebo and comparison of 5 mg to placebo in ACR20 had to be statistically significant; Least squares mean difference = -0.34, 95% CI 2-sided [-0.73 to 0.04], Standard Error of Mean 0.20

3. Primary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Month 3
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom, arise, eat, walk, reach, grip, hygiene and common activities over past week. Each item scored on 4-point scale, 0 to 3: 0=no difficulty; 1=some difficulty;2=much difficulty; 3=unable to do. Overall score was computed as sum of domain sc ores and divided by number of domains answered. Total possible score range 0-3: 0=least difficulty and 3=extreme difficulty. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 3 analysis.
Time Frame: Baseline, Month 3
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 315 | 309 | 156
units on a scale
  Baseline | 1.41 (0.68) | 1.39 (0.66) | 1.31 (0.68)
  Change at Month 3 | -0.3 (0.45) | -0.4 (0.48) | -0.1 (0.38)
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Change at Month 3: Least squares mean difference and corresponding 95% confidence interval (CI) was calculated using a mixed-effect repeated measure model with treatment, visit and treatment-by-visit interaction as fixed effect and participant as random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For comparison of 10 mg to placebo to be statistically significant in this measure, comparison of 10 mg to placebo in mTSS had to be significant; Least squares mean difference = -0.40, 95% CI 2-sided [-0.49 to -0.31], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; Change at Month 3: Least squares mean difference and corresponding 95% CI was calculated using a mixed-effect repeated measure model with treatment, visit and treatment-by-visit interaction as fixed effect and participant as random effect; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For comparison of 5 mg to placebo to be statistically significant, comparison of 10 mg to placebo and comparison of 5 mg to placebo in mTSS had to be statistically significant; Least squares mean difference = -0.25, 95% CI 2-sided [-0.34 to -0.16], Standard Error of Mean 0.05

4. Primary Outcome: Percentage of Participant With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 at Month 6
Description: DAS28-4 (ESR) calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joint count, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) less than or equal to (=<) 3.2 implied low disease activity, greater than (>) 3.2 to 5.1 implied moderate to high disease activity and less than (<) 2.6=remission. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 6 analysis.
Time Frame: Month 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Missing values due to withdrawal or advancement to active treatment before Month 6 were imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 265 | 257 | 129
percentage of participants | 7.17 | 15.95 | 1.55
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation to the binomial distribution was used to test the superiority of CP-690,550 10 mg to placebo and two-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal approximation — A step-down procedure was used to control for multiple comparisons. For comparison of 10 mg to placebo to be statistically significant in this measure, comparison of 10 mg to placebo in HAQ-DI had to be significant; Percent difference = 14.40, 95% CI 2-sided [9.44 to 19.36]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0034, Normal approximation — A step-down procedure was used to control for multiple comparisons. For comparison of 5 mg to placebo to be statistically significant, comparison of 10 mg to placebo and comparison of 5 mg to placebo in HAQ-DI had to be statistically significant; Percent difference = 5.61, 95% CI 2-sided [1.85 to 9.38]

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) at Month 1 and 3
Description: ACR20 response: >=20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Month 1, 3
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 309 | 309 | 154
percentage of participants
  Month 1 | 41.42 | 52.10 | 16.34
  Month 3 | 56.31 | 66.34 | 27.27

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 5
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: FAS population. 'N' (number of participants analyzed)signifies those participants who were evaluable for this measure. Missing values due to withdrawal or advancement to active treatment before Month 6 were imputed using NRI method. Data for time points after Month 12 shall be reported after completion of the end-of-study analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 309 | 309 | 79 | 75
percentage of participants
  Month 9 | 47.90 | 62.46 | 32.91 | 29.33
  Month 12 | 48.54 | 56.96 | 30.38 | 33.33

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) at Month 1, 3 and 6
Description: ACR50 response: greater than or equal to >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Month 1, 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. 'N' (number of participants analyzed)signifies those participants who were evaluable for this measure. Missing values due to withdrawal or advancement to active treatment before Month 6 were imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 309 | 309 | 154
percentage of participants
  Month 1 | 16.83 | 18.45 | 1.31
  Month 3 | 28.80 | 36.25 | 7.79
  Month 6 | 32.36 | 43.69 | 8.44

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 7
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction from baseline in both swollen and tender joint counts from baseline, received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 24. At Month 6, remaining participants received CP-690,550 5 mg or 10 mg tablet orally twice daily up to Month 24.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo
Number analyzed (Participants) | 309 | 309 | 79 | 75
percentage of participants
  Month 9 | 32.69 | 44.01 | 22.78 | 20.00
  Month 12 | 32.69 | 41.10 | 21.52 | 16.00

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) at Month 1, 3 and 6
Description: ACR70 response: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Month 1, 3, 6
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 309 | 309 | 154
percentage of participants
  Month 1 | 3.88 | 3.56 | 0.00
  Month 3 | 10.68 | 17.15 | 2.60
  Month 6 | 14.56 | 22.33 | 1.30

10. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 9
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 309 | 309 | 79 | 75
percentage of participants
  Month 9 | 18.45 | 28.48 | 8.86 | 12.00
  Month 12 | 18.77 | 27.51 | 10.13 | 12.00

11. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Baseline, Month 1, 3 and 6
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 316 | 309 | 156
units on a scale
  Baseline (n=316,309,156) | 5.22 (0.88) | 5.20 (0.87) | 5.16 (0.87)
  Month 1 (n=309,308,152) | 4.04 (1.14) | 3.84 (1.09) | 4.73 (1.10)
  Month 3 (n=294,299,145) | 3.62 (1.13) | 3.29 (1.14) | 4.54 (1.18)
  Month 6 (n=283,285,62) | 3.33 (1.12) | 2.96 (1.09) | 3.79 (1.06)

12. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Month 9, 12, 15, 18, 21 and 24
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 indicated low disease activity, >3.2 to 5.1 indicated moderate to high disease activity and <2.6 = remission.
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Data for time points after Month 12 will be reported after completion of the end-of-study analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 265 | 278 | 69 | 63
units on a scale
  Month 9 | 3.11 (1.17) | 2.88 (1.20) | 2.99 (1.11) | 3.03 (1.06)
  Month 12 | 3.07 (1.23) | 2.75 (1.14) | 3.05 (1.18) | 2.91 (1.05)

13. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Baseline, Month 1, 3 and 6
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, ESR (mm/hour) and PGA of disease activity (participant rated arthritis activity assessment with transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 316 | 306 | 154
units on a scale
  Baseline (n=316,306,154) | 6.34 (0.97) | 6.25 (0.99) | 6.27 (1.01)
  Month 1 (n=258,250,127) | 5.12 (1.32) | 4.84 (1.28) | 5.83 (1.17)
  Month 3 (n=249,248,122) | 4.58 (1.29) | 4.19 (1.34) | 5.57 (1.23)
  Month 6 (n=239,236,49) | 4.34 (1.24) | 3.90 (1.31) | 4.81 (1.21)

14. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Month 9, 12, 15, 18, 21 and 24
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, ESR (mm/hour) and PtGA of disease activity (participant rated arthritis activity assessment with transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 227 | 229 | 56 | 54
units on a scale
  Month 9 | 4.12 (1.26) | 3.84 (1.35) | 4.04 (1.33) | 3.87 (1.30)
  Month 12 | 4.09 (1.31) | 3.79 (1.34) | 4.20 (1.41) | 3.84 (1.35)

15. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP])
Description: DAS28-4 (CRP) was calculated from SJC and TJC using the 28 joints count, CRP [mg/L] and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 [CRP] <=3.2 implied low disease activity, DAS28-4 [CRP] >3.2 to 5.1 implied moderate to high disease activity and DAS28 <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6, 9, 12, 15, 18, 21, 24
Population: Since DAS28-4 (CRP) was determined to provide no new information over DAS28-4 (ESR) and DAS28-3 (CRP), there was a change in planned analysis and data was not analyzed for DAS28-4 (CRP).
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (3 Variables) (DAS28-3 [ESR])
Description: DAS28-3 (ESR) was calculated from the number of SJC and TJC using the 28 joints count and ESR (mm/hr). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (ESR) <=3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6, 9, 12, 15, 18, 21, 24
Population: Since DAS28-3 (ESR) was determined to provide no new information over DAS28-4 (ESR) and DAS28-3 (CRP), there was a change in planned analysis and data was not analyzed for DAS28-3 (ESR).
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Modified Total Sharp Scores (mTSS) at Baseline
Description: mTSS = sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline
Population: FAS included all randomized participants who received at least 1 dose of study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 286 | 295 | 139
units on a scale | 31.1 (47.71) | 37.3 (54.10) | 32.6 (41.80)

18. Secondary Outcome: Modified Total Sharp Scores (mTSS) at Month 12 and 24
Description: as for outcome 17
Time Frame: Month 12, 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Data for Month 24 will be reported after completion of the end-of-study analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 286 | 295 | 71 | 68
units on a scale | 31.4 (47.88) | 37.3 (54.03) | 36.1 (43.59) | 30.9 (41.18)

19. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Baseline, Month 1, 3 and 6
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0=least difficulty and 3=extreme difficulty.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 315 | 309 | 156
units on a scale
  Baseline (n=315,309,156) | 1.41 (0.68) | 1.39 (0.66) | 1.31 (0.68)
  Month 1 (n=309,308,153) | 1.16 (0.67) | 1.02 (0.65) | 1.25 (0.67)
  Month 3 (n=295,300,146) | 1.00 (0.65) | 0.84 (0.65) | 1.19 (0.69)
  Month 6 (n=283,285,62) | 0.94 (0.62) | 0.79 (0.64) | 1.09 (0.62)

20. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 19
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 265 | 278 | 69 | 63
units on a scale
  Month 9 | 0.91 (0.65) | 0.75 (0.64) | 0.95 (0.66) | 0.74 (0.67)
  Month 12 | 0.90 (0.65) | 0.76 (0.68) | 0.84 (0.66) | 0.74 (0.68)

21. Secondary Outcome: Patient Assessment of Arthritis Pain at Baseline, Month 1, 3 and 6
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) visual analogue scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 316 | 309 | 156
mm
  Baseline (n=316,309,156) | 58.39 (23.08) | 57.62 (24.10) | 55.01 (23.87)
  Month 1 (n=309,308,153) | 41.61 (24.08) | 33.91 (22.30) | 49.22 (24.51)
  Month 3 (n=295,300,146) | 34.47 (23.49) | 29.23 (21.95) | 46.96 (24.02)
  Month 6 (n=283,285,62) | 32.79 (22.90) | 29.05 (22.71) | 36.76 (22.14)

22. Secondary Outcome: Patient Assessment of Arthritis Pain at Month 9, 12, 15, 18, 21 and 24
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm visual analogue scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 265 | 278 | 69 | 63
mm
  Month 9 | 31.59 (23.13) | 27.14 (23.10) | 31.74 (23.26) | 27.54 (23.12)
  Month 12 | 30.54 (23.00) | 27.45 (24.56) | 27.99 (23.55) | 29.41 (26.22)

23. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Baseline, Month 1, 3, and 6
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS where 0 = very well and 100 = very poorly.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 316 | 308 | 156
mm
  Baseline (n=316,308,156) | 58.06 (23.62) | 56.45 (22.96) | 54.11 (22.87)
  Month 1 (n=309,308,153) | 41.26 (23.69) | 34.95 (21.43) | 48.30 (24.47)
  Month 3 (n=295,300,146) | 35.07 (22.68) | 29.11 (20.54) | 46.96 (24.09)
  Month 6 (n=283,285,62) | 33.48 (22.39) | 29.03 (22.68) | 38.87 (23.17)

24. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 23
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 265 | 278 | 69 | 63
mm
  Month 9 | 31.19 (22.10) | 28.05 (22.46) | 31.46 (23.22) | 27.41 (23.22)
  Month 12 | 31.77 (22.55) | 29.12 (24.06) | 29.60 (23.15) | 28.11 (24.09)

25. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis at Baseline, Month 1, 3 and 6
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 316 | 309 | 156
mm
  Baseline (n=316,309,156) | 59.44 (15.87) | 58.42 (17.08) | 55.90 (17.37)
  Month 1 (n=309,308,152) | 37.97 (18.58) | 35.19 (19.29) | 45.50 (19.57)
  Month 3 (n=294,300,146) | 30.12 (18.61) | 24.47 (17.51) | 43.29 (22.25)
  Month 6 (n=283,284,61) | 25.47 (18.62) | 20.44 (15.75) | 26.61 (17.73)

26. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 25
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 264 | 278 | 69 | 62
mm
  Month 9 | 21.68 (16.14) | 18.90 (15.89) | 19.92 (17.59) | 19.29 (15.53)
  Month 12 | 20.40 (15.71) | 17.97 (15.08) | 20.42 (16.63) | 18.79 (15.42)

27. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Baseline, Month 1, 3 and 6
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and is reported as 2 summary scores; physical component score and mental component score. Total score range for the summary scores = 0-100, where higher score represents higher level of functioning.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 315 | 309 | 156
units on a scale
  Baseline:physical functioning(n=315,309,156) | 32.16 (9.98) | 32.61 (9.86) | 33.50 (10.70)
  Baseline:role physical(n=315,309,156) | 34.61 (9.40) | 35.41 (9.73) | 36.69 (10.54)
  Baseline:social functioning(n=315,309,156) | 37.16 (11.05) | 39.17 (11.42) | 39.37 (11.54)
  Baseline:bodily pain(n=315,309,156) | 34.01 (7.52) | 34.64 (7.89) | 35.57 (8.05)
  Baseline:mental health(n=315,309,156) | 39.94 (11.30) | 40.45 (11.15) | 42.03 (11.28)
  Baseline:role emotional(n=315,309,156) | 35.64 (12.67) | 36.25 (13.37) | 37.43 (13.82)
  Baseline:vitality(n=315,309,156) | 40.62 (9.90) | 42.53 (9.67) | 42.97 (9.95)
  Baseline:general health(n=315,309,156) | 35.16 (9.07) | 36.03 (8.79) | 36.82 (8.11)
  Baseline:mental component(n=315,309,156) | 41.01 (11.54) | 42.24 (11.52) | 43.21 (11.90)
  Baseline:physical component(n=315,309,156) | 33.05 (7.94) | 33.75 (7.77) | 34.51 (8.03)
  Month 1:physical functioning(n=308,308,153) | 34.61 (9.96) | 36.72 (10.01) | 35.27 (10.48)
  Month 1:role physical(n=307,308,153) | 39.21 (10.04) | 41.02 (9.81) | 38.30 (10.24)
  Month 1:social functioning(n=308,308,153) | 41.70 (10.44) | 43.54 (10.06) | 41.01 (11.57)
  Month 1:bodily pain(n=308,308,153) | 39.75 (8.08) | 42.02 (8.41) | 37.31 (8.93)
  Month 1:mental health(n=308,308,153) | 43.70 (11.76) | 44.88 (10.82) | 42.70 (11.98)
  Month 1:role emotional(n=307,308,153) | 39.06 (12.34) | 41.13 (12.03) | 38.53 (12.47)
  Month 1:vitality(n=308,308,153) | 45.33 (10.33) | 46.84 (9.77) | 43.82 (10.40)
  Month 1:general health(n=308,308,153) | 38.49 (9.28) | 39.91 (9.00) | 37.70 (8.85)
  Month 1:mental component(n=307,308,153) | 44.90 (11.74) | 46.28 (10.70) | 43.86 (11.90)
  Month 1:physical component(n=307,308,153) | 36.99 (8.24) | 38.96 (8.07) | 36.25 (8.24)
  Month 3:physical functioning(n=295,300,146) | 36.40 (10.51) | 39.34 (10.66) | 35.39 (10.66)
  Month 3:role physical(n=295,300,146) | 39.83 (10.11) | 42.82 (9.98) | 38.37 (10.65)
  Month 3:social functioning(n=295,300,146) | 42.73 (10.60) | 44.50 (10.27) | 40.86 (11.23)
  Month 3:bodily pain(n=295,300,146) | 41.30 (9.23) | 44.43 (9.02) | 38.17 (9.16)
  Month 3:mental health(n=295,300,146) | 43.84 (11.82) | 45.52 (10.50) | 42.80 (11.47)
  Month 3:role emotional(n=295,300,146) | 39.52 (12.64) | 43.12 (11.97) | 38.20 (13.46)
  Month 3:vitality(n=295,300,146) | 46.72 (10.31) | 48.60 (9.52) | 44.24 (10.15)
  Month 3:general health(n=294,300,146) | 39.76 (9.31) | 41.20 (8.84) | 38.24 (8.79)
  Month 3:mental component(n=294,300,146) | 45.22 (11.69) | 47.05 (10.27) | 43.70 (11.68)
  Month 3:physical component(n=294,300,146) | 38.65 (8.62) | 41.30 (8.49) | 36.79 (8.39)
  Month 6:physical functioning(n=283,284,62) | 37.33 (10.51) | 39.76 (10.71) | 37.60 (8.70)
  Month 6:role physical(n=282,284,62) | 41.46 (10.16) | 43.37 (9.62) | 41.38 (8.78)
  Month 6:social functioning(n=283,285,62) | 42.99 (10.58) | 44.87 (10.53) | 42.79 (9.48)
  Month 6:bodily pain(n=283,285,62) | 41.90 (8.81) | 44.18 (9.37) | 40.70 (8.06)
  Month 6:mental health(n=283,285,62) | 44.46 (11.86) | 45.60 (11.34) | 43.37 (8.46)
  Month 6:role emotional(n=282,284,62) | 40.58 (12.54) | 42.71 (11.69) | 41.88 (10.80)
  Month 6:vitality(n=283,285,62) | 46.58 (10.11) | 48.52 (9.42) | 46.31 (9.14)
  Month 6:general health(n=283,285,62) | 40.40 (9.14) | 41.78 (9.24) | 39.90 (7.03)
  Month 6:mental component(n=282,284,62) | 45.39 (11.86) | 46.82 (10.85) | 45.42 (9.35)
  Month 6:physical component(n=282,284,62) | 39.69 (8.39) | 41.78 (8.56) | 39.21 (6.99)

28. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 27
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo, Then CP-690,550 5 mg: Placebo matched to CP-690,550 tablet orally twice daily for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction from baseline in both swollen and tender joint counts, received CP-690,550 5 mg tablet orally twice daily up to Month 24. At Month 6, remaining participants received CP-690,550 5 mg tablet orally twice daily up to Month 24.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 264 | 278 | 69 | 63
units on a scale
  Month 9:physical functioning | 37.94 (10.38) | 40.66 (10.70) | 38.31 (10.62) | 41.29 (11.80)
  Month 9:role physical | 41.41 (10.30) | 43.96 (9.86) | 41.48 (9.87) | 44.96 (10.21)
  Month 9:social functioning | 44.16 (10.13) | 45.20 (10.67) | 43.70 (10.10) | 45.90 (11.40)
  Month 9:bodily pain | 42.24 (8.90) | 44.17 (9.45) | 43.88 (8.56) | 47.17 (9.99)
  Month 9:mental health | 45.02 (11.18) | 45.05 (11.75) | 44.52 (11.29) | 48.35 (11.68)
  Month 9:role emotional | 41.66 (12.56) | 43.01 (11.72) | 41.85 (11.43) | 45.28 (11.54)
  Month 9:vitality | 47.50 (10.28) | 47.94 (9.81) | 46.23 (10.02) | 50.10 (9.83)
  Month 9:general health | 40.61 (9.16) | 42.02 (9.57) | 40.79 (8.64) | 43.98 (9.96)
  Month 9:mental component | 46.53 (11.50) | 46.38 (11.16) | 45.70 (11.01) | 49.07 (10.98)
  Month 9:physical component | 39.79 (8.38) | 42.49 (8.75) | 40.52 (8.47) | 43.44 (10.11)
  Month 12:physical functioning | 38.42 (10.83) | 40.01 (11.03) | 39.43 (10.51) | 42.27 (11.02)
  Month 12:role physical | 41.37 (10.19) | 43.59 (9.93) | 42.31 (10.62) | 45.15 (10.12)
  Month 12:social functioning | 43.48 (10.56) | 45.18 (10.54) | 44.28 (10.48) | 47.18 (10.29)
  Month 12:bodily pain | 42.83 (8.85) | 44.18 (9.59) | 43.60 (8.21) | 45.78 (9.89)
  Month 12:mental health | 44.73 (10.78) | 45.07 (11.22) | 44.66 (12.07) | 46.81 (11.48)
  Month 12:role emotional | 41.09 (12.73) | 42.80 (11.44) | 41.27 (12.59) | 44.38 (12.34)
  Month 12:vitality | 47.54 (10.15) | 48.12 (9.96) | 47.08 (11.04) | 49.20 (10.33)
  Month 12:general health | 40.35 (9.31) | 41.65 (9.38) | 40.48 (9.38) | 43.83 (9.53)
  Month 12:mental component | 45.82 (11.23) | 46.49 (10.61) | 45.55 (12.12) | 47.95 (10.79)
  Month 12:physical component | 40.23 (8.61) | 42.02 (8.82) | 41.22 (8.29) | 43.92 (9.20)

29. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline, Month 1, 3 and 6
Description: Participant-rated 12 item questionnaire to assess constructs of sleep over past week.7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range:0-100); sleep quantity(range:0-24), optimal sleep(yes or no). 9 item index measures of sleep disturbance provide composite scores: sleep problem summary, overall sleep problem. Except Adequacy, Optimal, Quantity of sleep, higher scores=more impairment. Scores transformed(actual raw score(RS) minus lowest possible score divided by possible RS range*100);total score range:0-100,higher score=more intensity of attribute.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 314 | 309 | 156
units on a scale
  Baseline:overall sleep problem(n=314,309,156) | 40.19 (20.12) | 39.70 (19.48) | 37.30 (18.32)
  Baseline:sleep problem summary(n=314,309,156) | 38.65 (20.70) | 38.47 (19.62) | 36.39 (18.50)
  Baseline:somnolence(n=314,309,156) | 36.75 (22.74) | 34.63 (22.05) | 33.72 (21.13)
  Baseline:snoring(n=312,309,156) | 34.36 (32.74) | 29.71 (31.28) | 29.36 (27.02)
  Baseline:quantity(n=315,308,155) | 6.46 (1.44) | 6.42 (1.41) | 6.46 (1.39)
  Baseline:sleep disturbance(n=314,309,156) | 41.04 (27.04) | 40.60 (26.64) | 36.49 (26.76)
  Baseline:awaken short of breath(n=314,309,156) | 17.90 (25.82) | 15.15 (23.60) | 14.74 (21.80)
  Baseline:adequacy(n=314,309,156) | 46.66 (28.23) | 45.83 (27.37) | 46.92 (26.14)
  Month 1:overall sleep problem(n=307,307,151) | 34.74 (20.68) | 33.90 (18.55) | 35.80 (19.12)
  Month 1:sleep problem summary(n=307,307,151) | 33.55 (20.86) | 33.33 (18.97) | 35.36 (19.46)
  Month 1:somnolence(n=307,307,151) | 32.18 (21.27) | 30.38 (20.22) | 32.80 (23.78)
  Month 1:snoring(n=308,306,151) | 31.36 (31.13) | 30.20 (31.25) | 29.80 (28.92)
  Month 1:quantity(n=307,306,153) | 6.60 (1.51) | 6.69 (1.31) | 6.38 (1.46)
  Month 1:sleep disturbance(n=308,307,151) | 34.04 (27.26) | 33.07 (24.86) | 33.73 (26.06)
  Month 1:awaken short of breath(n=308,307,151) | 15.26 (24.95) | 11.60 (19.70) | 14.97 (23.80)
  Month 1:adequacy(n=308,307,151) | 51.23 (28.31) | 49.61 (27.28) | 47.48 (26.79)
  Month 3:overall sleep problem(n=295,300,146) | 34.67 (20.37) | 34.10 (19.56) | 35.45 (18.16)
  Month 3:sleep problem summary(n=295,300,146) | 33.49 (20.90) | 33.30 (19.97) | 35.16 (19.04)
  Month 3:somnolence(n=295,300,146) | 31.86 (21.52) | 28.64 (20.43) | 32.65 (22.57)
  Month 3:snoring(n=295,299,146) | 33.49 (31.36) | 28.90 (29.81) | 30.27 (30.01)
  Month 3:quantity(n=295,300,146) | 6.69 (1.51) | 6.67 (1.34) | 6.59 (1.43)
  Month 3:sleep disturbance(n=295,300,146) | 34.43 (26.15) | 34.32 (26.81) | 33.15 (25.49)
  Month 3:awaken short of breath(n=295,300,146) | 16.61 (24.68) | 14.13 (21.52) | 15.75 (22.56)
  Month 3:adequacy(n=295,300,146) | 52.88 (29.21) | 50.93 (27.31) | 48.84 (25.74)
  Month 6:overall sleep problem(n=282,285,62) | 33.10 (19.14) | 32.67 (18.56) | 32.40 (13.97)
  Month 6:sleep problem summary(n=282,285,62) | 32.67 (20.38) | 32.07 (18.84) | 31.56 (15.05)
  Month 6:somnolence(n=283,285,62) | 30.60 (21.25) | 28.16 (20.17) | 27.74 (18.31)
  Month 6:snoring(n=283,285,62) | 31.87 (29.85) | 31.51 (30.29) | 29.03 (29.12)
  Month 6:quantity(n=283,285,62) | 6.66 (1.46) | 6.66 (1.41) | 6.65 (1.32)
  Month 6:sleep disturbance(n=282,285,62) | 31.76 (23.72) | 32.10 (24.14) | 31.61 (21.56)
  Month 6:awaken short of breath(n=283,285,62) | 15.90 (25.21) | 13.47 (21.19) | 13.23 (20.47)
  Month 6:adequacy(n=283,285,62) | 53.14 (27.54) | 52.32 (26.99) | 51.77 (26.64)

30. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline, Month 1, 3 and 6
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Number of participants with optimal sleep are reported.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 315 | 309 | 156
participants
  Baseline (n=315,309,156) | 140 | 132 | 70
  Month 1 (n=309,309,153) | 144 | 156 | 67
  Month 3 (n=295,300,146) | 140 | 150 | 71
  Month 6 (n=283,285,139) | 132 | 140 | 64

31. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) at Month 12, 18 and 24
Description: as for outcome 29
Time Frame: Month 12, 18, 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 248 | 264 | 67 | 63
units on a scale
  Month 12:overall sleep problem | 32.50 (18.21) | 32.68 (19.05) | 30.92 (17.24) | 28.34 (17.87)
  Month 12:sleep problem summary | 31.69 (18.69) | 31.97 (19.21) | 31.69 (18.18) | 28.73 (17.96)
  Month 12:somnolence | 30.53 (20.71) | 29.75 (21.78) | 28.96 (20.81) | 25.40 (18.62)
  Month 12:snoring | 31.77 (30.75) | 30.91 (31.14) | 31.64 (30.18) | 25.71 (25.25)
  Month 12:quantity | 6.73 (1.20) | 6.67 (1.26) | 6.73 (1.46) | 6.71 (1.52)
  Month 12:sleep disturbance | 30.72 (23.45) | 31.43 (24.09) | 29.35 (23.07) | 24.01 (24.02)
  Month 12:awaken short of breath | 14.19 (22.23) | 13.48 (20.86) | 15.82 (20.16) | 13.33 (22.14)
  Month 12:adequacy | 53.35 (27.11) | 52.16 (26.33) | 55.37 (25.66) | 53.02 (28.77)

32. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Month 12, 18 and 24
Description: as for outcome 30
Time Frame: Month 12, 18, 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Data reported for Month 12. For time points after Month 12, data will be reported after completion of the end-of-study analysis.
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 251 | 265 | 67 | 63
participants | 131 | 134 | 36 | 28

33. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Baseline, Month 1, 3, and 6
Description: FACIT-Fatigue is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 315 | 307 | 155
units on a scale
  Baseline (n=315,307,155) | 28.59 (10.62) | 29.49 (10.62) | 31.07 (11.06)
  Month 1 (n=309,306,150) | 33.13 (10.47) | 34.31 (10.19) | 31.52 (10.63)
  Month 3 (n=295,300,146) | 34.19 (10.29) | 36.14 (9.53) | 31.51 (11.10)
  Month 6 (n=283,284,61) | 34.36 (9.95) | 36.47 (9.76) | 33.69 (9.06)

34. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Month 12, 18 and 24
Description: as for outcome 33
Time Frame: Month 12, 18, 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 250 | 265 | 67 | 62
units on a scale | 35.06 (10.00) | 35.88 (10.04) | 35.58 (10.65) | 37.29 (9.98)

35. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score at Baseline, Month 3 and 6
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 313 | 309 | 153
units on a scale
  Baseline (n=313,309,153) | 0.43 (0.31) | 0.47 (0.31) | 0.47 (0.30)
  Month 3 (n=261,262,125) | 0.60 (0.27) | 0.67 (0.22) | 0.52 (0.30)
  Month 6 (n=283,285,62) | 0.62 (0.25) | 0.69 (0.23) | 0.59 (0.24)

36. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score at Month 12, 18 and 24
Description: as for outcome 35
Time Frame: Month 12, 18, 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 251 | 265 | 67 | 63
units on a scale | 0.64 (0.25) | 0.69 (0.26) | 0.63 (0.30) | 0.74 (0.22)

37. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Baseline, Month 3 and 6
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (5-items); Physical Demands scale (6-item); Mental-Interpersonal Demands Scale (9-items); Output Demands scale (5-items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). Work Loss Index, which represented percentage of lost work over time period relative to a normative population, was derived (total score:0[no loss] to 100[complete loss of work]).
Time Frame: Baseline, Month 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 155 | 157 | 87
units on a scale
  Baseline:time management(n=147,146,81) | 49.74 (25.59) | 41.93 (26.90) | 44.02 (28.39)
  Baseline:physical demands(n=149,152,86) | 50.17 (24.18) | 50.11 (24.19) | 49.96 (26.67)
  Baseline:mental demands(n=151,151,86) | 33.91 (25.41) | 29.28 (24.47) | 33.13 (27.93)
  Baseline:output demands(n=149,147,83) | 38.81 (26.66) | 36.85 (25.95) | 40.57 (29.38)
  Baseline:work loss index(n=155,157,87) | 11.13 (5.71) | 9.98 (5.66) | 10.99 (6.78)
  Month 3:time management(n=107,116,52) | 45.18 (31.06) | 35.87 (33.78) | 41.11 (27.36)
  Month 3:physical demands(n=106,124,55) | 47.11 (29.37) | 44.06 (32.26) | 46.02 (25.36)
  Month 3:mental demands(n=111,124,55 | 27.92 (27.18) | 23.52 (27.09) | 34.24 (27.87)
  Month 3:output demands(n=108,119,54) | 32.71 (27.67) | 25.48 (28.69) | 39.23 (28.44)
  Month 3:work loss index(n=111,127,55) | 9.77 (6.29) | 7.86 (6.44) | 10.89 (6.40)
  Month 6:time management(n=97,116,19) | 37.90 (30.57) | 34.33 (33.47) | 40.53 (32.70)
  Month 6:physical demands(n=104,116,19) | 48.00 (29.47) | 43.01 (34.57) | 43.90 (31.26)
  Month 6:mental demands(n=103,117,18) | 25.30 (29.75) | 21.95 (28.40) | 32.43 (30.69)
  Month 6:output demands(n=101,117,18) | 29.43 (29.61) | 24.26 (29.30) | 35.56 (26.78)
  Month 6:work loss index(n=105,123,19) | 8.78 (6.75) | 7.47 (6.57) | 10.05 (6.54)

38. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Month 12, 18 and 24
Description: as for outcome 37
Time Frame: Month 12, 18, 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively. Data for time points after Month 12 will be reported after completion of the end-of-study analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 94 | 118 | 23 | 33
units on a scale
  Month 12:time management(n=92,108,22,32) | 35.82 (31.75) | 31.30 (31.68) | 43.69 (32.76) | 37.58 (36.88)
  Month 12:physical demands(n=91,110,22,33) | 45.64 (33.67) | 46.16 (33.53) | 47.01 (32.96) | 41.10 (35.89)
  Month 12:mental demands(n=93,115,23,33) | 21.24 (25.05) | 20.42 (25.99) | 39.29 (35.39) | 27.70 (33.57)
  Month 12:output demands(n=93,107,23,31) | 23.71 (26.59) | 21.18 (26.52) | 37.12 (34.59) | 33.67 (34.78)
  Month 12:work loss index(n=94,118,23,33) | 7.78 (5.94) | 6.88 (5.98) | 11.33 (7.64) | 9.24 (7.91)

39. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Baseline, Month 3 and 6
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost: visit to doctor, non-medical practitioner, nursing home, hospital, surgery, emergency room(ER) treatment, diagnostic tests, over-night stay, home healthcare services, aids/devices used. Indirect costs associated with functional disability: employment status, willingness to work, work disability due to RA, sick leave, part time work, ability to perform chores, chores done by family, friends or housekeeper. Assessment was based on 0 to 2-point scale; higher score=higher medical cost.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 315 | 306 | 155
units on a scale
  Baseline: Seen any doctor (n=315, 305, 154) | 1.14 (0.34) | 1.15 (0.36) | 1.16 (0.36)
  Baseline:Treated in emergency room(n=315,306,155) | 1.93 (0.26) | 1.96 (0.19) | 1.94 (0.23)
  Baseline:Admitted for overnight stay (n=22,12,9) | 0.27 (0.63) | 0.25 (0.45) | 0.00 (0.00)
  Baseline:Hospitalization(n=315,306,155) | 1.94 (0.23) | 1.94 (0.24) | 1.97 (0.18)
  Baseline:Outpatient surgery(n=315,305,155) | 1.97 (0.16) | 1.96 (0.20) | 1.97 (0.18)
  Baseline:Non-study diagnostic test(n=315,306,155) | 1.82 (0.39) | 1.83 (0.37) | 1.85 (0.36)
  Baseline:In nursing home(n=315,306,155) | 1.99 (0.10) | 1.99 (0.10) | 1.99 (0.11)
  Baseline:Home healthcare services(n=315,306,154) | 1.97 (0.16) | 1.99 (0.10) | 1.98 (0.14)
  Baseline:Required aids/devices(n=315,306,155) | 1.87 (0.34) | 1.91 (0.29) | 1.90 (0.30)
  Baseline:Non-medical practitioner(n=315,306,155) | 1.97 (0.18) | 1.94 (0.23) | 1.95 (0.21)
  Baseline:Currently employed(n=314,306,155) | 1.65 (0.48) | 1.60 (0.49) | 1.62 (0.49)
  Baseline:Feel well enough to work(n=182,166,89) | 1.87 (0.33) | 1.86 (0.35) | 1.82 (0.39)
  Baseline:Unable to work due to RA(n=185,169,88) | 1.37 (0.48) | 1.37 (0.48) | 1.32 (0.47)
  Baseline:Lost job/retired early(n=184,169,86) | 1.61 (0.49) | 1.61 (0.49) | 1.67 (0.47)
  Baseline:Work disabled due to RA(n=186,168,88) | 1.52 (0.50) | 1.61 (0.49) | 1.52 (0.50)
  Baseline:Retired(n=193,171,92) | 1.51 (0.50) | 1.51 (0.50) | 1.52 (0.50)
  Baseline:Sick leave due to RA(n=236,236,123) | 1.83 (0.38) | 1.81 (0.39) | 1.76 (0.43)
  Baseline:Performed part time work(n=235,236,121) | 1.87 (0.34) | 1.87 (0.33) | 1.90 (0.30)
  Baseline:Performed paid work(n=235,235,122) | 1.60 (0.49) | 1.62 (0.49) | 1.61 (0.49)
  Baseline:Unable to do chores(n=312,302,152) | 1.38 (0.48) | 1.43 (0.50) | 1.43 (0.50)
  Baseline:Chores by housekeeper(n=315,305,155) | 1.83 (0.37) | 1.85 (0.36) | 1.90 (0.30)
  Baseline:Chores by family/friends(n=315,305,155) | 1.49 (0.50) | 1.50 (0.50) | 1.53 (0.50)
  Month 3:Seen any doctor(n=259,260,121) | 1.31 (0.46) | 1.31 (0.46) | 1.28 (0.45)
  Month 3:Treated in emergency room(n=259,260,121) | 1.95 (0.23) | 1.95 (0.22) | 1.97 (0.18)
  Month 3:Admitted for overnight stay (n=14,12,4) | 0.64 (0.84) | 0.08 (0.29) | 0.00 (0.00)
  Month 3:Hospitalization(n=259,260,121) | 1.97 (0.18) | 1.98 (0.12) | 1.99 (0.09)
  Month 3:Outpatient surgery(n=259,260,121) | 1.97 (0.17) | 1.98 (0.12) | 1.99 (0.09)
  Month 3:Non-study diagnostic test(n=259,260,121) | 1.86 (0.35) | 1.83 (0.37) | 1.88 (0.32)
  Month 3:In nursing home(n=259,260,121) | 2.00 (0.00) | 2.00 (0.06) | 2.00 (0.00)
  Month 3:Home healthcare services(n=257,260,121) | 1.98 (0.14) | 2.00 (0.06) | 2.00 (0.00)
  Month 3:Required aids/devices(n=259,260,121) | 1.91 (0.29) | 1.91 (0.29) | 1.89 (0.31)
  Month 3:Non-medical practitioner(n=259,260,121) | 1.98 (0.14) | 1.97 (0.17) | 1.98 (0.16)
  Month 3:Currently employed(n=259,260,121) | 1.63 (0.48) | 1.57 (0.50) | 1.60 (0.49)
  Month 3:Feel well enough to work(n=147,140,68) | 1.78 (0.41) | 1.73 (0.45) | 1.82 (0.38)
  Month 3:Unable to work due to RA(n=148,139,67) | 1.44 (0.50) | 1.50 (0.50) | 1.39 (0.49)
  Month 3:Lost job/retired early(n=148,139,67) | 1.64 (0.48) | 1.63 (0.49) | 1.57 (0.50)
  Month 3:Work disabled due to RA(n=150,140,68) | 1.53 (0.50) | 1.64 (0.48) | 1.57 (0.50)
  Month 3:Retired(n=150,142,70) | 1.51 (0.50) | 1.42 (0.50) | 1.63 (0.49)
  Month 3:Sick leave due to RA(n=175,200,89) | 1.89 (0.31) | 1.93 (0.26) | 1.82 (0.39)
  Month 3:Performed part time work(n=176,196,89) | 1.91 (0.29) | 1.94 (0.24) | 1.87 (0.34)
  Month 3:Performed paid work(n=174,197,88) | 1.70 (0.46) | 1.76 (0.43) | 1.69 (0.46)
  Month 3:Unable to do chores(n=257,256,121) | 1.60 (0.49) | 1.70 (0.46) | 1.52 (0.50)
  Month 3:Chores by housekeeper(n=257,259,121) | 1.90 (0.30) | 1.92 (0.27) | 1.90 (0.30)
  Month 3:Chores by family/friends(n=257,259,121) | 1.67 (0.47) | 1.73 (0.44) | 1.53 (0.50)
  Month 6:Seen any doctor(n=282,285,61) | 1.21 (0.41) | 1.21 (0.41) | 1.31 (0.47)
  Month 6:Treated in emergency room(n=283,285,61) | 1.94 (0.23) | 1.96 (0.20) | 1.93 (0.25)
  Month 6:Admitted for overnight stay (n=17,12,4) | 0.12 (0.33) | 0.00 (0.00) | 1.00 (0.15)
  Month 6:Hospitalization(n=283,285,61) | 1.99 (0.10) | 1.99 (0.10) | 1.93 (0.25)
  Month 6:Outpatient surgery(n=283,285,61) | 1.96 (0.20) | 1.99 (0.10) | 1.95 (0.22)
  Month 6:Non-study diagnostic test(n=282,284,61) | 1.79 (0.41) | 1.85 (0.36) | 1.82 (0.39)
  Month 6:In nursing home(n=283,285,61) | 1.99 (0.10) | 2.00 (0.00) | 2.00 (0.00)
  Month 6:Home healthcare services(n=282,284,61) | 1.98 (0.13) | 1.99 (0.08) | 1.98 (0.13)
  Month 6:Required aids/devices(n=283,285,61) | 1.90 (0.30) | 1.94 (0.24) | 1.97 (0.18)
  Month 6:Non-medical practitioner(n=283,285,61) | 1.98 (0.14) | 1.97 (0.17) | 1.97 (0.18)
  Month 6:Currently employed(n=283,285,61) | 1.65 (0.48) | 1.59 (0.49) | 1.70 (0.46)
  Month 6:Feel well enough to work(n=176,154,38) | 1.77 (0.42) | 1.73 (0.44) | 1.79 (0.41)
  Month 6:Unable to work due to RA(n=177,155,40) | 1.47 (0.50) | 1.55 (0.50) | 1.43 (0.50)
  Month 6:Lost job/retired early(n=173,158,38) | 1.69 (0.46) | 1.63 (0.49) | 1.79 (0.41)
  Month 6:Work disabled due to RA(n=174,154,38) | 1.52 (0.50) | 1.66 (0.48) | 1.66 (0.48)
  Month 6:Retired(n=178,157,41) | 1.49 (0.50) | 1.48 (0.50) | 1.61 (0.49)
  Month 6:Sick leave due to RA(n=195,216,37) | 1.92 (0.27) | 1.95 (0.22) | 1.89 (0.31)
  Month 6:Performed part time work(n=193,215,37) | 1.96 (0.20) | 1.94 (0.23) | 1.92 (0.28)
  Month 6:Performed paid work(n=193,216,37) | 1.76 (0.43) | 1.76 (0.43) | 1.65 (0.48)
  Month 6:Unable to do chores(n=281,284,61) | 1.63 (0.48) | 1.80 (0.40) | 1.64 (0.48)
  Month 6:Chores by housekeeper(n=281,285,61) | 1.89 (0.31) | 1.92 (0.28) | 1.90 (0.30)
  Month 6:Chores by family/friends(n=281,285,61) | 1.70 (0.46) | 1.76 (0.42) | 1.75 (0.43)

40. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Month 12, 18 and 24
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost:visit to doctor,non-medical practitioner,nursing home,hospital,surgery,emergency room(ER) treatment,diagnostic tests, over-night stay,home healthcare services, aids/devices used. Indirect costs associated with functional disability:employment status,willingness to work,work disability due to RA,sick leave,part time work,ability to perform chores,chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale;higher score=higher medical cost.
Time Frame: Month 12, 18, 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively. Data for time points after Month 12 shall be reported after completion of the end-of-study analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 250 | 265 | 67 | 63
units on a scale
  Month 12:Seen any doctor(n=250,265,67,63) | 1.21 (0.41) | 1.18 (0.39) | 1.16 (0.37) | 1.17 (0.38)
  Month 12:Treated in ER(n=250,265,67,63) | 1.93 (0.26) | 1.96 (0.20) | 1.94 (0.24) | 1.95 (0.21)
  Month 12:Admitted for overnight stay(n=18,11,4,3) | 0.17 (0.38) | 0.18 (0.40) | 0.25 (0.50) | 0.33 (0.58)
  Month 12:Hospitalization(n=250,265,67,63) | 1.97 (0.18) | 1.98 (0.12) | 1.97 (0.17) | 1.98 (0.13)
  Month 12:Outpatient surgery(n=250,265,67,63) | 1.95 (0.22) | 1.98 (0.12) | 1.99 (0.12) | 1.98 (0.13)
  Month 12:Diagnostic test(n=250,265,67,63) | 1.79 (0.41) | 1.81 (0.39) | 1.87 (0.34) | 1.86 (0.35)
  Month 12:In nursing home(n=250,265,67,63) | 1.99 (0.09) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00)
  Month 12:Home healthcare services(n=249,264,67,63) | 1.99 (0.09) | 2.00 (0.06) | 2.00 (0.00) | 2.00 (0.00)
  Month 12:Required aids/devices(n=250,265,67,63) | 1.90 (0.31) | 1.94 (0.23) | 1.94 (0.24) | 1.98 (0.13)
  Month 12:Non-medical practitioner(n=250,265,67,63) | 1.98 (0.13) | 1.98 (0.15) | 1.94 (0.24) | 1.98 (0.13)
  Month 12:Currently employed(n=250,265,67,63) | 1.62 (0.49) | 1.57 (0.50) | 1.66 (0.48) | 1.51 (0.50)
  Month 12:Feel well enough to work(n=151,141,41,29) | 1.73 (0.45) | 1.65 (0.48) | 1.80 (0.40) | 1.62 (0.49)
  Month 12:Unable to work due to RA(n=150,141,41,29) | 1.50 (0.50) | 1.53 (0.50) | 1.49 (0.51) | 1.66 (0.48)
  Month 12:Lost job/retired early(n=151,143,41,29) | 1.73 (0.45) | 1.69 (0.47) | 1.68 (0.47) | 1.83 (0.38)
  Month 12:Work disabled due to RA(n=151,143,42,30) | 1.60 (0.49) | 1.66 (0.47) | 1.57 (0.50) | 1.77 (0.43)
  Month 12:Retired(n=154,140,42,30) | 1.51 (0.50) | 1.44 (0.50) | 1.52 (0.51) | 1.57 (0.50)
  Month 12:Sick leave due to RA(n=168,200,46,48) | 1.93 (0.25) | 1.93 (0.26) | 1.98 (0.15) | 1.90 (0.31)
  Month 12:Performed part time work(n=167,199,46,48) | 1.99 (0.11) | 1.96 (0.18) | 2.00 (0.00) | 1.94 (0.24)
  Month 12:Performed paid work(n=168,200,46,48) | 1.77 (0.42) | 1.81 (0.39) | 1.78 (0.42) | 1.75 (0.44)
  Month 12:Unable to do chores(n=246,265,67,63) | 1.65 (0.48) | 1.78 (0.42) | 1.82 (0.39) | 1.75 (0.44)
  Month 12:Chores by housekeeper(n=249,264,67,63) | 1.92 (0.27) | 1.93 (0.25) | 1.94 (0.24) | 2.00 (0.00)
  Month 12:Chores by family/friends(n=249,264,67,63) | 1.75 (0.44) | 1.79 (0.41) | 1.76 (0.43) | 1.79 (0.41)

41. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA/non-RA related number of events including visits to doctor, non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 273 | 262 | 132
events
  Baseline:Doctor visit(n=273,262,132) | 3.78 (4.24) | 4.00 (5.07) | 4.80 (5.61)
  Baseline:RA related doctor visit(n=271,262,131) | 1.16 (0.70) | 1.20 (0.80) | 1.25 (0.67)
  Baseline:Hospital ER visit(n=19,11,9) | 1.42 (0.77) | 1.73 (1.27) | 1.22 (0.67)
  Baseline:RA related ER visit(n=23,12,9) | 0.74 (0.81) | 0.83 (1.34) | 0.56 (0.73)
  Baseline:Hospitalization(n=18,18,5) | 1.17 (0.51) | 1.17 (0.38) | 1.00 (0.00)
  Baseline:RA related hospitalization(n=18,19,5) | 1.11 (0.58) | 1.32 (1.34) | 1.40 (0.55)
  Baseline:Outpatient surgery(n=8,13,5) | 1.13 (0.35) | 1.85 (2.76) | 1.00 (0.00)
  Baseline:RA related outpatient surgery(n=8,14,5) | 0.38 (0.52) | 0.43 (0.85) | 0.40 (0.55)
  Baseline:Non-study diagnostic test(n=56,51,22) | 1.80 (1.18) | 1.67 (1.16) | 1.73 (1.12)
  Baseline:RA related diagnostic test(n=57,53,23) | 0.74 (1.09) | 0.77 (1.19) | 0.83 (1.15)
  Baseline:Non-medical practitioner visit(n=10,17,7) | 12.50 (12.29) | 10.88 (13.09) | 12.57 (13.23)
  Baseline:RA related non-medical visit(n=11,18,7) | 1.00 (0.77) | 1.00 (0.84) | 1.57 (1.27)
  Month 3:Doctor visit(n=181,181,89) | 2.85 (1.79) | 3.08 (2.76) | 3.27 (3.73)
  Month 3:RA related doctor visit(n=181,180,89) | 0.92 (0.63) | 0.79 (0.54) | 0.87 (0.61)
  Month 3:Hospital ER visit(n=14,11,4) | 1.29 (0.61) | 1.45 (0.93) | 1.00 (0.00)
  Month 3:RA related ER visit(n=14,13,4) | 0.29 (0.73) | 0.15 (0.55) | 0.00 (0.00)
  Month 3:Hospitalization(n=9,4,1) | 1.00 (0.00) | 1.25 (0.50) | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:RA related hospitalization(n=9,4,1) | 0.11 (0.33) | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:Outpatient surgery(n=8,5,1) | 1.25 (0.46) | 1.20 (0.45) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:RA related outpatient surgery(n=8,5,1) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:Non-study diagnostic test(n=32,43,13) | 1.41 (0.71) | 1.56 (1.35) | 1.46 (0.97)
  Month 3:RA related diagnostic test(n=37,44,14) | 0.14 (0.35) | 0.07 (0.25) | 0.14 (0.36)
  Month 3:Non-medical practitioner visit(n=4,8,3) | 7.50 (11.03) | 3.63 (1.51) | 22.33 (11.24)
  Month 3:RA related non-medical visit(n=4,8,3) | 0.50 (1.00) | 0.38 (0.52) | 0.67 (0.58)
  Month 6:Doctor visit(n=226,225,43) | 3.00 (2.89) | 2.72 (2.28) | 4.51 (6.05)
  Month 6:RA related doctor visit(n=225,224,43) | 0.87 (0.56) | 0.86 (0.56) | 0.91 (0.61)
  Month 6:Hospital ER visit(n=15,12,4) | 1.27 (0.59) | 1.33 (0.49) | 2.25 (2.50)
  Month 6:RA related ER visit(n=16,12,4) | 0.25 (0.58) | 0.33 (0.78) | 0.50 (1.00)
  Month 6:Hospitalization(n=3,3,4) | 1.00 (0.00) | 1.00 (0.00) | 1.25 (0.50)
  Month 6:RA related hospitalization(n=3,3,4) | 0.33 (0.58) | 0.33 (0.58) | 0.50 (1.00)
  Month 6:Outpatient surgery(n=12,2,3) | 1.33 (0.89) | 1.00 (0.00) | 1.00 (0.00)
  Month 6:RA related outpatient surgery(n=12,3,3) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Month 6:Non-study diagnostic test(n=58,41,11) | 1.78 (1.83) | 1.73 (1.40) | 2.00 (1.00)
  Month 6:RA related diagnostic test(n=60,44,11) | 0.25 (0.68) | 0.25 (0.69) | 0.09 (0.30)
  Month 6:Non-medical practitioner visit(n=6,8,2) | 15.00 (17.34) | 6.13 (4.55) | 25.00 (7.07)
  Month 6:RA related non-medical visit(n=6,8,3) | 1.50 (1.52) | 0.25 (0.46) | 1.67 (0.58)

42. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Month 12, 18 and 24
Description: as for outcome 41
Time Frame: Month 12, 18, 24
Population: FAS. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points for each group respectively. Data for time points after Month 12 will be reported after completion of the end-of-study analysis.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 197 | 221 | 56 | 52
events
  Month 12:Doctor visit(n=197,221,56,52) | 2.70 (2.74) | 2.43 (2.26) | 3.27 (4.02) | 2.81 (3.91)
  Month 12:RA related doctor visit (n=197,220,56,52) | 0.92 (0.52) | 0.89 (0.43) | 0.93 (0.60) | 0.88 (0.47)
  Month 12:Hospital ER visit(n=18,11,4,3) | 1.61 (1.58) | 1.00 (0.00) | 1.25 (0.50) | 1.00 (0.00)
  Month 12:RA related ER visit(n=18,11,4,3) | 0.11 (0.32) | 0.09 (0.30) | 0.25 (0.50) | 0.00 (0.00)
  Month 12:Hospitalization(n=8,4,2,1) | 1.00 (0.00) | 1.00 (0.00) | 1.50 (0.71) | 1.00 (0.00)
  Month 12:RA related hospitalization(n=8,4,2,1) | 0.50 (0.76) | 0.50 (0.58) | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 12:Outpatient surgery(n=13,4,1,1) | 2.31 (2.39) | 1.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 12:RA related outpatient surgery(n=13,4,1,1) | 0.46 (0.66) | 0.25 (0.50) | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 12:Non-study diagnostic test(n=50,47,9,8) | 1.98 (1.49) | 1.55 (1.14) | 2.00 (1.00) | 1.88 (0.83)
  Month 12:RA related diagnostic test(n=52,50,9,9) | 0.27 (0.56) | 0.24 (0.48) | 0.22 (0.67) | 0.11 (0.33)
  Month 12:Non-medical practitioner visit(n=4,6,4,1) | 12.00 (5.86) | 9.83 (15.03) | 10.00 (7.12) | 9.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 12:RA related non-medical visit(n=4,6,4,1) | 1.25 (0.96) | 0.17 (0.41) | 0.75 (0.96) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.

43. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains.Any RA or non-RA related number of days spent in hospital, nursing home, aids/devices used, on sick leave, work per week, performed part time work, performed paid work, chores done by housekeeper and chores done by family/friends.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 158 | 152 | 73
days
  Baseline:Hospital length of stay(n=18,18,5) | 10.94 (9.12) | 20.22 (19.70) | 22.20 (15.37)
  Baseline:Days in nursing home(n=3,3,2) | 14.33 (12.10) | 17.67 (3.51) | 15.50 (7.78)
  Baseline:Days aids/devices used(n=41,25,14) | 109.63 (108.88) | 74.08 (66.11) | 102.21 (75.87)
  Baseline:RA related aids used(n=42,29,14) | 1.93 (1.24) | 1.59 (1.02) | 1.64 (0.50)
  Baseline:Days of work per week(n=109,121,59) | 5.01 (1.14) | 5.14 (0.92) | 4.93 (1.39)
  Baseline:Days on sick leave due to RA(n=41,44,29) | 13.17 (21.61) | 16.84 (27.67) | 15.45 (25.69)
  Baseline:Days of part time work(n=30,29,12) | 9.07 (12.62) | 12.07 (16.50) | 26.92 (32.20)
  Baseline:Paid work, bothered by RA(n=92,88,48) | 29.13 (30.81) | 31.59 (30.12) | 31.90 (31.61)
  Baseline:Chores by housekeeper(n=50,44,15) | 19.06 (23.91) | 20.89 (33.69) | 17.87 (18.71)
  Baseline:Chores by family(n=158,152,73) | 36.28 (34.40) | 30.39 (34.00) | 37.11 (34.99)
  Month 3:Hospital length of stay(n=9,4,1) | 5.67 (4.95) | 16.25 (26.51) | 32.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:Days in nursing home(n=0,1,0) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 28.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 3:Days aids/devices used(n=23,22,13) | 107.22 (102.77) | 69.36 (60.36) | 85.00 (57.64)
  Month 3:RA related aids used(n=23,24,14) | 1.78 (1.04) | 1.21 (0.51) | 1.21 (0.70)
  Month 3:Days of work per week(n=97,113,48) | 5.03 (1.03) | 5.25 (0.92) | 4.88 (1.21)
  Month 3:Days on sick leave due to RA(n=19,15,16) | 12.16 (20.51) | 8.20 (19.95) | 11.13 (21.56)
  Month 3:Days of part time work(n=16,12,12) | 9.44 (11.51) | 9.42 (13.17) | 15.67 (26.60)
  Month 3:Paid work, bothered by RA(n=52,48,27) | 20.60 (27.99) | 17.42 (21.52) | 34.59 (33.28)
  Month 3:Chores by housekeeper(n=25,21,12) | 17.00 (20.88) | 6.05 (33.69) | 21.75 (18.71)
  Month 3:Chores by family(n=84,70,57) | 31.37 (34.32) | 21.46 (29.48) | 27.53 (33.51)
  Month 6:Hospital length of stay(n=3,3,4) | 12.67 (9.07) | 8.33 (6.66) | 9.25 (2.50)
  Month 6:Days in nursing home(n=3,0,0) | 24.00 (3.61) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 6:Days aids/devices used(n=27,17,2) | 93.44 (104.39) | 87.12 (61.54) | 110.00 (98.99)
  Month 6:RA related aids used(n=28,18,2) | 1.36 (1.06) | 1.56 (1.20) | 2.00 (0.00)
  Month 6:Days of work per week(n=98,117,18) | 5.02 (1.16) | 5.29 (0.78) | 4.94 (1.00)
  Month 6:Days on sick leave due to RA(n=15,11,4) | 14.93 (24.05) | 14.18 (25.86) | 24.25 (43.84)
  Month 6:Days of part time work(n=8,12,3) | 11.88 (14.99) | 11.33 (11.44) | 4.33 (1.15)
  Month 6:Paid work, bothered by RA(n=46,52,13) | 18.87 (25.75) | 18.67 (19.85) | 12.85 (15.66)
  Month 6:Chores by housekeeper(n=30,24,6) | 15.90 (22.43) | 18.08 (26.29) | 44.00 (40.99)
  Month 6:Chores by family(n=85,66,15) | 29.41 (33.22) | 29.65 (33.02) | 34.87 (40.65)

44. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Month 12, 18 and 24
Description: as for outcome 43
Time Frame: Month 12, 18, 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 94 | 114 | 23 | 31
days
  Month 12:Hospital length of stay(n=8,4,2,1) | 10.13 (6.58) | 7.00 (5.35) | 2.50 (2.12) | 3.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 12:Days in nursing home(n=2,0,0,0) | 11.50 (2.12) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 12:Days aids/devices used(n=25,14,4,1) | 85.68 (95.83) | 138.21 (110.42) | 100.50 (57.63) | 180.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 12:RA related aids used(n=26,16,4,1) | 1.62 (1.06) | 1.94 (1.69) | 1.00 (0.82) | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 12:Days of work per week(n=94,114,23,31) | 5.01 (1.15) | 5.20 (0.75) | 4.65 (1.15) | 4.87 (1.26)
  Month 12:Days on sick leave due to RA(n=11,15,1,5) | 32.27 (39.24) | 5.13 (4.42) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 5.60 (4.51)
  Month 12:Days of part time work(n=3,7,0,3) | 16.33 (17.90) | 15.57 (21.19) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 31.67 (51.39)
  Month 12:Paid work, bothered by RA(n=38,38,10,12) | 20.89 (24.78) | 18.58 (24.28) | 23.80 (28.35) | 28.17 (35.51)
  Month 12:Chores by housekeeper(n=18,18,4,0) | 14.06 (20.23) | 10.11 (11.20) | 24.50 (43.68) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 12:Chores by family(n=62,56,16,13) | 30.15 (33.03) | 23.77 (31.80) | 38.38 (39.32) | 16.77 (24.59)

45. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home healthcare services, chores done by housekeeper, chores done by family or friends, work done and work missed were reported.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 158 | 152 | 71
hours per day
  Baseline:Home healthcare services(n=6,2,3) | 1.50 (0.84) | 3.00 (1.41) | 1.33 (0.58)
  Baseline:RA related home HC services(n=8,4,3) | 1.00 (0.76) | 1.50 (1.00) | 0.67 (1.15)
  Baseline:Work done(n=108,121,59) | 8.01 (4.05) | 8.22 (4.41) | 8.12 (5.25)
  Baseline:Missed work due to RA(n=30,30,12) | 7.03 (9.98) | 5.33 (4.47) | 4.33 (6.29)
  Baseline:Chores by housekeeper(n=51,44,14) | 4.27 (2.19) | 4.98 (2.76) | 4.21 (2.22)
  Baseline:Chores by family(n=158,152,71) | 3.95 (4.33) | 3.66 (3.87) | 3.49 (4.16)
  Month 3:Home healthcare services(n=5,1,0) | 1.20 (0.45) | 4.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 3:RA related home HC services(n=5,1,0) | 0.80 (0.84) | 3.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 3:Work done(n=97,113,48) | 7.71 (4.83) | 8.25 (3.60) | 7.42 (2.47)
  Month 3:Missed work due to RA(n=16,12,12) | 9.94 (16.85) | 3.17 (2.92) | 5.42 (6.16)
  Month 3:Chores by housekeeper(n=25,21,12) | 4.84 (4.59) | 4.48 (2.18) | 4.83 (2.62)
  Month 3:Chores by family(n=83,70,56) | 4.31 (9.29) | 3.64 (4.73) | 4.04 (4.45)
  Month 6:Home healthcare services(n=5,2,1) | 2.20 (2.17) | 3.00 (2.83) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 6:RA related home HC services(n=5,2,1) | 1.20 (0.84) | 1.50 (2.12) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 6:Work done(n=98,117,18) | 8.15 (4.15) | 7.90 (1.85) | 7.56 (3.05)
  Month 6:Missed work due to RA(n=8,12,3) | 2.38 (1.60) | 2.50 (1.62) | 1.00 (1.73)
  Month 6:Chores by housekeeper(n=30,23,6) | 4.97 (3.00) | 4.87 (2.32) | 2.67 (1.21)
  Month 6:Chores by family(n=83,67,15) | 3.13 (2.39) | 3.25 (4.09) | 2.93 (1.79)

46. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Month 12, 18 and 24
Description: as for outcome 45
Time Frame: Month 12, 18, 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 95 | 114 | 23 | 31
hours per day
  Month 12:Home healthcare services(n=2,1,0,0) | 20.50 (27.58) | 4.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 12:RA related home HC services(n=2,1,0,0) | 0.50 (0.71) | 3.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 12:Work done(n=95,114,23,31) | 7.78 (3.81) | 7.92 (1.88) | 7.48 (2.02) | 8.03 (2.09)
  Month 12:Missed work due to RA(n=3,7,0,3) | 1.33 (1.15) | 8.71 (12.42) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 2.67 (1.53)
  Month 12:Chores by housekeeper(n=17,17,4,0) | 4.47 (2.27) | 4.53 (1.70) | 5.25 (3.40) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 12:Chores by family(n=62,56,16,13) | 3.31 (2.36) | 3.20 (2.16) | 3.75 (2.38) | 2.31 (0.95)

47. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: Work performance of participants on number of days bothered was based on a 0 to 10-point scale, where higher score indicated lower work performance.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 204 | 202 | 104
units on a scale
  Baseline (n=204,202,104) | 5.29 (3.09) | 4.88 (3.03) | 4.68 (3.03)
  Month 3 (n=151,176,81) | 3.81 (3.11) | 3.11 (2.67) | 4.40 (2.87)
  Month 6 (n=160,185,29) | 3.73 (3.18) | 2.99 (2.94) | 3.41 (2.85)

48. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Month 12, 18 and 24
Description: as for outcome 47
Time Frame: Month 12, 18, 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Data for time points after Month 12 shall be reported after completion of the end-of-study analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 144 | 163 | 39 | 44
units on a scale | 3.19 (3.13) | 2.66 (2.80) | 2.51 (2.54) | 2.66 (2.72)

49. Other Pre Specified Outcome: Percentage of Participants With Sustained American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: >=20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP. Participants with sustained ACR20 response for 2, 3, 4 and 5 consecutive visits were analyzed up to Month 12.
Time Frame: Baseline through Month 12, Month 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Data up to Month 12 reported. For time period after Month 12, data will be reported after completion of the end-of-study analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 316 | 309 | 79 | 75
percentage of participants
  2 consecutive visits | 16.8 | 13.9 | 21.5 | 16.9
  3 consecutive visits | 13.0 | 14.2 | 27.8 | 28.6
  4 consecutive visits | 16.5 | 16.2 | 11.4 | 10.4
  5 consecutive visits | 18.7 | 33.7 | 7.6 | 3.9

50. Other Pre Specified Outcome: Percentage of Participants With Sustained American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP. Participants with sustained ACR50 response for 2, 3, 4 and 5 consecutive visits were analyzed up to Month 12.
Time Frame: Baseline through Month 12, Month 24
Population: FAS population: all randomized participants who received at least 1 dose of study medication. Data up to Month 12 reported. For time period after Month 12, data will be reported after completion of the end-of-study analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 316 | 309 | 79 | 77
percentage of participants
  2 consecutive visits | 12.0 | 16.5 | 21.5 | 19.5
  3 consecutive visits | 7.9 | 11.3 | 13.9 | 13.0
  4 consecutive visits | 8.2 | 12.3 | 0.0 | 2.6
  5 consecutive visits | 7.3 | 9.4 | 1.3 | 0.0

51. Other Pre Specified Outcome: Percentage of Participants With Sustained American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP. Participants with sustained ACR70 response for 2, 3, 4 and 5 consecutive visits were analyzed up to Month 12.
Time Frame: Baseline through Month 12, Month 24
Population: as for outcome 50
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 316 | 309 | 79 | 77
percentage of participants
  2 consecutive visits | 6.6 | 10.4 | 8.9 | 18.2
  3 consecutive visits | 4.1 | 6.8 | 5.1 | 2.6
  4 consecutive visits | 2.8 | 7.1 | 0.0 | 0.0
  5 consecutive visits | 1.3 | 2.3 | 0.0 | 0.0

52. Other Pre Specified Outcome: Percentage of Participants With Sustained Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) Less Than 2.6
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission. Participants with sustained DAS28-3 (CRP) response less than 2.6 for 2, 3, 4 and 5 consecutive visits were analyzed up to Month 12.
Time Frame: Baseline through Month 12, Month 24
Population: as for outcome 49
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 316 | 309 | 79 | 75
percentage of participants
  2 consecutive visits | 13.0 | 12.6 | 19.0 | 18.2
  3 consecutive visits | 7.9 | 11.7 | 5.1 | 7.8
  4 consecutive visits | 5.7 | 13.3 | 3.8 | 0.0
  5 consecutive visits | 2.2 | 3.2 | 1.3 | 0.0

53. Other Pre Specified Outcome: Percentage of Participants With Sustained Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission. Participants with sustained DAS28-4 (ESR) response less than 2.6 for 2, 3, 4 and 5 consecutive visits were analyzed up to Month 12.
Time Frame: Baseline through Month 12, Month 24
Population: FAS population. Data up to Month 12 reported. For time period after Month 12, data will be reported after completion of the end-of-study analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 316 | 309 | 79 | 77
percentage of participants
  2 consecutive visits | 4.4 | 5.5 | 3.8 | 7.8
  3 consecutive visits | 1.0 | 3.6 | 1.3 | 1.3
  4 consecutive visits | 1.9 | 3.2 | 0.0 | 0.0
  5 consecutive visits | 0.0 | 1.0 | 0.0 | 0.0

54. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than or Equal to 3.2 at Month 1, 3 and 6
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joint count, ESR (mm/hour) and patient's global assessment (PtGA) of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Month 1, 3, 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 265 | 257 | 129
percentage of participants
  Month 1 | 6.98 | 10.40 | 3.15
  Month 3 | 13.96 | 25.29 | 3.88
  Month 6 | 14.34 | 28.40 | 3.10

55. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than or Equal to 3.2 at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 54
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Missing values due to withdrawal or advancement to active treatment before Month 6 were imputed using NRI method. Data for time points after Month 12 will be reported after completion of the end-of-study analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 265 | 257 | 65 | 64
percentage of participants
  Month 9 | 18.87 | 33.46 | 10.77 | 12.50
  Month 12 | 21.13 | 28.79 | 9.23 | 17.19

56. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 at Month 1, 3 and 6
Description: as for outcome 54
Time Frame: Month 1, 3, 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 265 | 257 | 129
percentage of participants
  Month 1 | 1.55 | 2.80 | 0.00
  Month 3 | 5.28 | 11.28 | 1.55
  Month 6 | 7.17 | 15.95 | 1.55

57. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 54
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 55
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 265 | 257 | 65 | 64
percentage of participants
  Month 9 | 10.57 | 14.01 | 4.62 | 3.13
  Month 12 | 9.81 | 14.40 | 3.08 | 7.81

58. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) Less Than or Equal to 3.2 at Month 1, 3 and 6
Description: as for outcome 11
Time Frame: Month 1, 3, 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 309 | 308 | 154
percentage of participants
  Month 1 | 23.62 | 31.49 | 6.58
  Month 3 | 35.28 | 44.48 | 11.69
  Month 6 | 37.86 | 50.97 | 10.39

59. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) Less Than or Equal to 3.2 at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 11
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 55
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 309 | 308 | 79 | 75
percentage of participants
  Month 9 | 38.51 | 52.27 | 25.32 | 24.00
  Month 12 | 40.13 | 51.95 | 24.05 | 24.00

60. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) Less Than 2.6 at Month 1, 3 and 6
Description: as for outcome 11
Time Frame: Month 1, 3, 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 309 | 308 | 154
percentage of participants
  Month 1 | 11.33 | 9.09 | 1.97
  Month 3 | 20.39 | 26.95 | 5.19
  Month 6 | 22.98 | 36.36 | 5.19

61. Other Pre Specified Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) Less Than 2.6 at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 11
Time Frame: Month 9, 12, 15, 18, 21, 24
Population: as for outcome 55
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 309 | 308 | 79 | 75
percentage of participants
  Month 9 | 26.86 | 38.31 | 22.78 | 14.67
  Month 12 | 28.80 | 39.61 | 17.72 | 18.67

62. Other Pre Specified Outcome: Association Between Genomic and Metabonomic Variation
Time Frame: Month 24
Reporting Status: Not Posted

63. Other Pre Specified Outcome: Change From Baseline in Blood Pressure (BP) at Month 1, 3 and 6
Description: BP: pressure exerted by the blood upon the walls of the blood vessels and especially arteries, usually measured on the radial artery using a sphygmomanometer. Systolic BP: the highest arterial blood pressure of a cardiac cycle occurring immediately after systole of the left ventricle of the heart. Diastolic BP: the lowest arterial blood pressure of a cardiac cycle occurring during diastole of the heart.
Time Frame: Baseline, Month 1, 3, 6
Population: Safety analysis set: all randomized participants who received at least 1 dose of study medication. 'N' (number of participants analyzed)=participants evaluable for the measure. 'n'=participants evaluable at given time points for each group respectively. Data for time points after Month 12 will be reported after completion of end-of-study analysis.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 316 | 309 | 156
millimeters of mercury (mmHg)
  Baseline:systolic BP(n=316,309,156) | 125.85 (13.23) | 123.95 (15.05) | 123.87 (14.32)
  Baseline:diastolic BP(n=316,309,156) | 77.27 (8.41) | 77.25 (9.34) | 76.81 (8.70)
  Change at Month 1:systolic BP(n=309,308,153) | -1.6 (11.87) | 0.5 (12.40) | 0.5 (11.96)
  Change at Month 1:diastolic BP(n=309,308,153) | -0.1 (8.06) | 0.1 (7.99) | 0.5 (7.19)
  Change at Month 3:systolic BP(n=295,299,146) | -1.2 (12.33) | 0.6 (13.55) | 0.7 (11.75)
  Change at Month 3:diastolic BP(n=295,299,146) | 1.0 (8.76) | 0.5 (8.61) | -0.0 (8.63)
  Change at Month 6:systolic BP(n=283,285,62) | -0.5 (13.57) | 1.1 (13.15) | -0.6 (11.63)
  Change at Month 6:diastolic BP(n=283,285,62) | 0.2 (8.63) | 0.8 (8.45) | -0.4 (7.74)

64. Other Pre Specified Outcome: Change From Baseline in Blood Pressure (BP) at Month 9, 12, 15, 18, 21 and 24
Description: as for outcome 63
Time Frame: Baseline, Month 9, 12, 15, 18, 21, 24
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 316 | 309 | 79 | 77
mmHg
  Baseline:systolic BP(n=316,309,79,77) | 125.83 (13.23) | 123.95 (15.05) | 124.37 (14.78) | 123.35 (13.90)
  Baseline:diastolic BP(n=316,309,79,77) | 77.27 (8.41) | 77.25 (9.34) | 77.11 (8.62) | 76.51 (8.81)
  Change at Month 9:systolic BP(n=265,278,69,63) | -0.4 (13.51) | 1.8 (14.21) | -1.1 (12.44) | 0.3 (13.09)
  Change at Month 9:diastolic BP(n=265,278,69,63) | 0.1 (8.92) | 1.3 (8.78) | -0.0 (7.96) | 1.0 (6.66)
  Change at Month 12:systolic BP(n=251,265,67,63) | -1.3 (13.93) | 1.1 (14.28) | 1.1 (10.91) | 1.3 (14.59)
  Change at Month 12:diastolic BP(n=251,265,67,63) | -0.9 (9.37) | 0.6 (8.94) | 1.8 (7.50) | 0.7 (9.32)

65. Other Pre Specified Outcome: Change From Baseline in Heart Rate at Month 1, 3, 6, 9, 12, 15, 18, 21 and 24
Time Frame: Baseline, Month 1, 3, 6, 9, 12, 15, 18, 21, 24
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings as per planned analysis but not statistically summarized.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

66. Other Pre Specified Outcome: Change From Baseline in Body Temperature at Month 1, 3, 6, 9, 12, 15, 18, 21 and 24
Time Frame: Baseline, Month 1, 3, 6, 9, 12, 15, 18, 21, 24
Population: as for outcome 65
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690,550 5 mg (Up To Month 3): Participants received CP-690,550 5 mg tablet orally twice daily up to Month 3.
- CP-690,550 10 mg (Up to Month 3): Participants received CP-690,550 10 mg tablet orally twice daily up to Month 3.
- Placebo (Up to Month 3): Participants received placebo matched to CP-690,550 tablet orally twice daily up to Month 3.
- CP-690,550 5 mg (Month 3 to 6): Participants who received either CP-690,550 5 mg or matching placebo up to Month 3, received CP-690,550 5 mg tablet orally twice daily from Month 3 to 6.
- CP-690,550 10 mg (Month 3 to 6): Participants who received either CP-690,550 10 mg or matching placebo up to Month 3, received CP-690,550 10 mg tablet orally twice daily from Month 3 to 6.
- Placebo (Month 3 to 6): Participants received placebo matched to CP-690,550 tablet orally twice daily from Month 3 to 6.
- CP-690,550 5 mg (Post Month 6): Participants who received either CP-690,550 5 mg or matching placebo up to Month 6, received CP-690,550 5 mg tablet orally twice daily from Month 6 to 24.
- CP-690,550 10 mg (Post Month 6): Participants who received either CP-690,550 10 mg or matching placebo up to Month 6, received CP-690,550 10 mg tablet orally twice daily from Month 6 to 24.
Arm/Group | CP-690,550 5 mg (Up To Month 3) | CP-690,550 10 mg (Up to Month 3) | Placebo (Up to Month 3) | CP-690,550 5 mg (Month 3 to 6) | CP-690,550 10 mg (Month 3 to 6) | Placebo (Month 3 to 6) | CP-690,550 5 mg (Post Month 6) | CP-690,550 10 mg (Post Month 6)
Serious Adverse Events (participants affected / at risk) | 12/321 | 10/316 | 5/160 | 18/363 | 8/353 | 5/81 | 14/402 | 13/395
Other Adverse Events (participants affected / at risk) | 70/321 | 49/316 | 21/160 | 33/363 | 27/353 | 4/81 | 66/402 | 79/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Up To Month 3) (N=321) | CP-690,550 10 mg (Up to Month 3) (N=316) | Placebo (Up to Month 3) (N=160) | CP-690,550 5 mg (Month 3 to 6) (N=363) | CP-690,550 10 mg (Month 3 to 6) (N=353) | Placebo (Month 3 to 6) (N=81) | CP-690,550 5 mg (Post Month 6) (N=402) | CP-690,550 10 mg (Post Month 6) (N=395)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Necrotising retinitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device breakage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug interaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colonoscopy (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian granulosa-theca cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infarction (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Up To Month 3) (N=321) | CP-690,550 10 mg (Up to Month 3) (N=316) | Placebo (Up to Month 3) (N=160) | CP-690,550 5 mg (Month 3 to 6) (N=363) | CP-690,550 10 mg (Month 3 to 6) (N=353) | Placebo (Month 3 to 6) (N=81) | CP-690,550 5 mg (Post Month 6) (N=402) | CP-690,550 10 mg (Post Month 6) (N=395)
Nausea (Gastrointestinal disorders) | 7 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 8 | 2 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 14 | 13 | 1 | 13 | 9 | 4 | 22 | 22
Upper respiratory tract infection (Infections and infestations) | 9 | 7 | 5 | 17 | 9 | 0 | 13 | 15
Urinary tract infection (Infections and infestations) | 9 | 3 | 4 | 0 | 0 | 0 | 10 | 17
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 3 | 9 | 0 | 9 | 10
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 5 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 18 | 4 | 3 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 11 | 4 | 1 | 0 | 0 | 0 | 8 | 6

LIMITATIONS AND CAVEATS:
Results include data of 1-year analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.